CLINICAL TRIAL: NCT04798833
Title: An Integrated Newborn Care Kit to Save Newborn Lives and Improve Health Outcomes in Gilgit-Baltistan, Pakistan
Brief Title: Newborn Care Kit to Save Lives in GB, Pakistan
Acronym: iNCK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Aga Khan Foundation (Other); Aga Khan Health Services (Other); Aga Khan University (Other)
Responsible Party: Principal Investigator, Shaun Morris, Clinician-Scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TTS181021048
Record Dates: First submitted 2021-03-09; First posted 2021-03-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Mortality; Omphalitis; Post-Partum Hemorrhage
Keywords: Neonatal Mortality; Neonatal kit; Pakistan; Randomized Control Trial; Chlorhexidine; Omphalitis; Newborn; Birth; Post-Partum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrated Newborn Care Kit (Experimental): The integrated newborn care kit will contain a clean birth kit to be used at the time of delivery either at home or in a facility, three misoprostol tablets (200ug each), 4% chlorhexidine solution, sunflower oil emollient, temperature monitoring strip or sticker, a fleece blanket, a reusable, non-electric, heating device, and a pictorial instruction guide. Lady Health Workers will be equipped with a hand-held electronic scale to identify low birth weight newborns.
  Participants in this arm will receive the same local standard of care as the no intervention arm.
  Interventions: Device: Integrated Newborn Care Kit (iNCK)
- Control (Local Standard of Care) (No Intervention): In the control arm, LHWs will deliver the local standard of care, which entails both anti-natal and post-natal LHW home visits. As part of standard practice, LHWs visit pregnant women in their homes during the 3rd trimester, at which time these health workers:
  * Provide instructions regarding proper nutrition during pregnancy
  * Encourage that delivery take place in a facility
  * Discuss the fundamentals of safe water, sanitation, and hygiene behavior
  * Encourage exclusive breastfeeding
  These community health workers will identify early danger signs in newborns such as infections and teach caregivers to identify the same symptoms, so that early interventions can be made. If danger signs are identified, the LHW will refer newborns to the appropriate level of health care.

INTERVENTIONS:
Device: Integrated Newborn Care Kit (iNCK) — Contents of the integrated newborn care kit:
  * Clean birth kit: sterile blade, clean plastic sheet, plastic gloves, hand soap, cord ties/clamp, maternity pad to absorb post-natal bleeding, 10 cotton balls for applying Chlorhexidine (CHX) to the umbilical stump.
  * 3x200 µg dissolvable tablets of misoprostol to be ingested prophylactically following delivery of the baby and before delivery of the placenta to prevent post-partum hemorrhage
  * 4% CHX solution (15 mL)
  * Sunflower oil emollient (50 mL)
  * Temperature monitoring strip or sticker
  * Fleece blanket for the newborn
  * Click to heat warmer
  * Pictorial guide that illustrates how and when to use each kit component
  * Handheld electronic scale with suspended cloth sling (the scale will not be included with the kit but rather one will be issued to each Lady Health Worker in the experimental arm)
  Other Names: Neonatal Care Kit
  Other Names: Neonatal Care Kit
  Arms: Integrated Newborn Care Kit

SUMMARY:
Neonatal deaths account for almost half of all deaths in children under 5 years of age. Pakistan has the world's highest neonatal mortality rate (NMR), and many of these deaths are preventable. In this study, the investigators propose the use of an evidence-based, integrated newborn care kit (iNCK) to promote safer delivery, provide early identification of danger signs, improve newborn health, and reduce NMR. The investigators hypothesize that use of the iNCK will result in at least a 25% reduction in NMR among participants who receive the iNCK compared with participants who do not receive the iNCK.

DETAILED DESCRIPTION:
While some progress has been made towards reducing global under-5 mortality, in 2019, an estimated 2.4 million newborn deaths still occurred worldwide, accounting for 47% of all under-five deaths. Most neonatal deaths are caused by prematurity, sepsis, and intrapartum-related complications.

Pakistan has the highest neonatal mortality rate (NMR) in the world, at 42 deaths per 1,000 live births. Gilgit-Baltistan (GB), Pakistan's remote, northern-most administrative territory, is afflicted with some of the country's worst NMRs. High rates of home deliveries, low adoption of safe birth practices, inadequate cord care, and high maternal mortality contribute to this health disparity. GB's geography, climate, and underdeveloped infrastructure also largely restrict access to health care facilities. Health care at the community level in Pakistan is primarily supported by the Lady Health Worker (LHW) Programme. LHWs form a cadre of government-supported community health workers who provide newborn and maternal health services in GB. However, each of these health care workers is responsible for approximately 1,000 people, which restricts both availability and comprehensiveness of care, particularly for families that live in hard to reach areas.

Many proven, cost-effective ways to save newborn lives and improve wellbeing exist; however, they are not always available to those who need them most, nor are they packaged into a single portable kit that can be used in the home. An easy-to-use kit consisting of low cost, evidence-based interventions has potential to improve health status, reduce NMR, and provide more timely access to health services in remote areas such as GB. Between April 2014 and August 2015, the investigators conducted a community-based, cluster randomized intervention trial examining the effectiveness of delivering an integrated newborn care kit (iNCK) to pregnant women in Rahim Yar Khan (RYK), Punjab, Pakistan. The iNCKs were delivered by LHWs, who also educated participants how to use the different kit components. Neonatal mortality and morbidity outcomes were compared between iNCK recipients and a local control group who received the same standard of care, but no iNCK. The investigators found that while distribution of the iNCK did not significantly reduce neonatal mortality, utilization of the iNCK significantly reduced the risk of omphalitis and fever. Moreover, using the LHW network to distribute the intervention proved a feasible delivery mechanism.

The findings from the RYK trial suggest that while a network of community health workers can reliably deliver integrated interventions to pregnant women, further investigation is needed to improve the integration of educational content and maximize the iNCK's potential health benefits. Moreover, effective delivery of maternal health interventions through the iNCK warrants examination, as Pakistan experiences some of the world's highest rates of maternal mortality, of which post-partum hemorrhage (PPH) is a leading cause.

ELIGIBILITY:
Inclusion Criteria:

* Resides in a village with LHW coverage in participating union councils (clusters) in Astore, Diamer, Shigar, Ghanche, Kharmang, and Skardu, districts of GB, Pakistan
* In their 3rd trimester of pregnancy (≥ week 27 gestational age)
* Intends to be present in the study catchment area between day 29 and 35 postnatal age
* Provides written informed consent or assent
* Starting in approximately month 26 of the study, only women ≥36 weeks of gestational age will be enrolled.

Exclusion Criteria:

* Does not reside within the study's catchment area at the time of enrolment
* Plans to relocate outside of the study catchment area within one month after the delivery of their newborn(s) and not return to the study catchment area
* Does not provide written informed consent or assent
* Lives in a village without LHW coverage

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27448 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
All-cause neonatal mortality | Day 29 postnatal age
  Death from any cause within the first 28 days of life

SECONDARY OUTCOMES:
Cumulative incidence of omphalitis | Day 29 postnatal age
  Cumulative incidence of omphalitis among neonates where omphalitis is defined as:
  1. redness around the base of the baby's umbilical stump or surrounding skin OR
  2. the presence of pus on or near the baby's umbilical stump
Cumulative incidence of post-partum hemorrhage (PPH) | Day 29 postnatal age
  Cumulative incidence of PPH is self-reported. PPH is defined as having experienced any of the following:
  1. Post-delivery vaginal bleeding that pooled on the mattress/floor where the delivery took place
  2. Having sought health care for post-delivery vaginal bleeding
  3. Having received a blood transfusion after delivery
  4. Having been diagnosed with PPH
  5. Vaginal bleeding being reported as the cause of the mother's death
Health facility utilization | Day 29 postnatal age
  Self-reported health facility utilization by pregnant women, and/or neonates and mothers in the first month post-partum
Cumulative incidence of hypothermia among participants in the experimental arm | Day 29 postnatal age
  Cumulative incidence of hypothermia defined by color change in temperature monitoring strip or sticker that indicates lower than normal temperature
Cumulative incidence of fever among participants in the experimental arm | Day 29 postnatal age
  Cumulative incidence of fever defined by color change in temperature monitoring strip or sticker that indicates higher than normal temperature
Correlates of iNCK instructional compliance | Day 29 postnatal age
  Correlates of iNCK instructional compliance, using a process analysis to explore the correlation between compliance and maternal, infant, sociodemographic characteristics, and Lady Health Worker teaching quality
Correlates of willingness to pay for the iNCK | 29 postnatal age
  Explore the correlation between maternal, infant, and sociodemographic characteristics, and knowledge, attitudes, practice, and willingness to pay for the iNCK
Cause-specific neonatal mortality | Day 29 postnatal age
  Death from specific causes within the first 28 days of life

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Morris, MD, MPH, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Pakistan (2):
  - Aga Khan Health Services, Pakistan, Islamabad
  - Aga Khan University, Karachi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fadaleh SMA, Pell LG, Yasin M, Farrar DS, Khan SH, Tanner Z, Paracha S, Madhani F, Bassani DG, Ahmed I, Soofi SB, Taljaard M, Spitzer RF, Bhutta ZA, Morris SK. An integrated newborn care kit (iNCK) to save newborn lives and improve health outcomes in Gilgit Baltistan (GB), Pakistan: study protocol for a cluster randomized controlled trial. BMC Public Health. 2023 Dec 11;23(1):2480. doi: 10.1186/s12889-023-17322-y. PMID 38082395